CLINICAL TRIAL: NCT01513213
Title: Correlation of PaCO2 to the Inspired and Expired Oxygen Gradient
Acronym: O2 Fraction
Status: Completed | Type: Observational
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 5119S-11
Record Dates: First submitted 2012-01-05; First posted 2012-01-20 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Neurosurgery
Keywords: Arterial cannulation; Blood gas; Carbon dioxide; Arterial blood; Oxygen; Oxygen fractions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate whether a correlation exists between the partial pressure of carbon dioxide existing within arterial blood and the gradient between inhaled and exhaled fractions of oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65.
* Scheduled for surgical procedure that will last at least 2 hours.
* Arterial cannulation is planned because of either the complexity of the surgery or patient comorbidity.
* At least two arterial blood gas analyses are planned during the surgery.

Exclusion Criteria:

* No arterial cannulation is necessary or planned for the procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults age 18 to 65 scheduled for a surgical procedure that will last at least two hours and for whom arterial cannulation and at least two arterial blood gas analyses are planned during the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Correlate the level of carbon dioxide within arterial blood to inspired and expired oxygen gradient. | At least 2 hours
  Compare the levels of carbon dioxide found in the patient's blood to the amounts of carbon dioxide and oxygen in the air that the patient inhales and exhales. If a relationship exists between the levels of carbon dioxide in the blood and the levels of carbon dioxide and oxygen inhaled and exhaled by the patient, anesthesiologists will be able to use this relationship to adjust ventilators during anesthesia without having to take blood from an artery.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur M Lam, MD, FRCPC, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States